CLINICAL TRIAL: NCT04100902
Title: The Effect of Allergen Immunotherapy on Anti-viral Immunity in Patients With Allergic Asthma - A Randomized, Double-blind, Placebo-controlled Trial of HDM-AIT
Brief Title: The Effect of Allergen Immunotherapy on Anti-viral Immunity in Patients With Allergic Asthma
Acronym: VITAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other); ALK-Abelló A/S (Industry); Lund University (Other)
Responsible Party: Principal Investigator, Celeste Porsbjerg, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VITAL
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Allergic Asthma Due to Dermatophagoides Pteronyssinus
Keywords: Allergic asthma; Allergen Immunotherapy; Anti-viral immunity; House dust mite

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Odactra 12-sq HDM sublingual tablet (Active Comparator): House Dust Mite, sublingual tablet
  Interventions: Drug: ODACTRA 12 SQ-HDM Sublingual Tablet
- Placebo sublingual tablet (Placebo Comparator): Placebo, sublingual tablet
  Interventions: Drug: Placebo sublingual tablet

INTERVENTIONS:
Drug: ODACTRA 12 SQ-HDM Sublingual Tablet — Subjects are randomized to either HDM-AIT or Placebo for 24 weeks of therapy
  Other Names: 12-SQ-HDM sublingual tablet
  Arms: Odactra 12-sq HDM sublingual tablet
Drug: Placebo sublingual tablet — Subjects are randomized to either HDM-AIT or Placebo for 24 weeks of therapy
  Arms: Placebo sublingual tablet

SUMMARY:
Aim: To investigate the possible immune modulatory effects of allergen immunotherapy (AIT) on respiratory immunity in patients with allergic asthma (AA).

Background: Allergic sensitization to aeroallergens is a common co-morbidity in asthma that is associated with more frequent and severe asthma attacks. The investigators have recently shown that patients with allergic asthma also have an increased risk of pneumonia, and hence allergy in asthma may be associated with a relative respiratory immunodeficiency. However, the increased risk was obliterated in patients treated with AIT.

Methods: Patients with asthma sensitized to house-dust mite (HDM) is enrolled in a randomized, double-blind, placebo-controlled study of HDM-AIT. Patients will be scheduled for 9 visits through 8 months including, randomization to 6 months of treatment with either HDM-AIT (Acarizax/Odactra) or placebo. Primary interferons (IFN) type I and III will be investigated in human bronchial epithelial cells as the primary outcome. Secondary outcomes such as: Inflammatory cytokines, immunologic phenotype and immunohistochemistry will be investigated in bronchial biopsies, blood, bronchoalveolar lavage fluid, sputum and HDM-patch biopsies as well as a thorough respiratory and allergic evaluation.

Expected outcomes: The investigators expect that, patients with AA have 1) decreased production of anti-viral type I and III IFN and that AIT increases these measures. 2) Anti-bacterial response is reduced through IL12, ß-defensin and IFN-γ and that AIT increases these measures. 3) Lastly, the investigators expect that T-cell response is dysregulated (Th1↓1/Th2↑) in patients with AA and that these findings are modulated in an immuno-protective direction after AIT.

Perspectives: This project will expand our understanding of the clinical significance of allergy in asthma in a completely novel direction and show how AIT may modulate the immune response to prevent infections.

DETAILED DESCRIPTION:
1.1 Background Respiratory viral infections are the major cause of acute worsening of asthma. Importantly too, these infections may also predispose to bacterial infections. Patients with allergic asthma suffer from more frequent lower respiratory tract infections, more severe and longer lasting lower respiratory tract symptoms compared to healthy controls. Hence, the need to use antibiotics may reflect in part the increased susceptibility to viral infection in allergic asthma. The investigators have recently demonstrated that patients with allergic asthma have an increased risk of being prescribed antibiotics for respiratory infections compared to non-allergic patients with asthma. Other studies have identified allergic sensitization and respiratory viral infections as synergetic risk factors in asthma exacerbations. These findings suggest a possible link between the allergic sensitization, asthma and an impaired immune response against respiratory infections. Furthermore, the investigators have found that allergen-specific immunotherapy (AIT) reduces the risk of being prescribed antibiotics for respiratory infections in patients with allergic asthma. These novel observations make it of interest to investigate mechanistic pathways in target cells subjected to AIT.

In a recent study, investigating potential mechanisms involved in the interaction between allergen and viral infection the investigators found that house dust mite (HDM) impairs viral stimulus (TLR3)-induced type I and type III interferons in bronchial epithelial cells from asthmatic patients and similarly in an in vivo mouse model of asthma exacerbation. This novel finding was accompanied with a direct effect of HDM on reducing TLR3 glycosylation. Hence, HDM exposure in patients with allergic asthma may also contribute to a defect antiviral response by interfering with components important for the anti-viral signalling such as TLR3. Furthermore, the investigators have observed that HDM has a capacity to induce over-expression of upstream Th2 cytokines such as IL-33, which may contribute to asthma exacerbations. In our studies HDM stands out amongst different allergens in causing both release of inflammatory inducing damage-associated metabolic patterns and impaired interferon response.

Inferentially, in this study the investigators will have the unique opportunity to examine effects of human in vivo HDM-AIT on the bronchial epithelial cell production of type I and type III interferons as well as the balance between Th1/and Th2 inflammation in response to viral and bacterial triggers. The investigators speculate that exposure to HDM-allergen may predispose to asthma exacerbations by causing dysregulation of the anti-viral interferon system as well as Th1/and Th2 inflammation and then that desensitization of patients with HDM-sensitive allergic asthma (AA) increases innate interferon response.

1.2 Hypothesis

1. Viral induced type I and type III IFN is increased in HBECS from patients with allergic asthma sensitized to HDM, after 24 weeks of Acarizax.
2. Viral induced type I and III IFN response is impaired in HBECs from patients with allergic asthma sensitized to HDM, before 24 weeks of Acarizax.

1.3 Investigational Medical Product (IMP): ACARIZAX Acarizax is sublingual allergen immunotherapy (SLIT) for the treatment of HDM allergic rhinitis (AR) and allergic asthma (AA). Acarizax is composed of standardized allergen extract from the HDMs' Dermatophagoides pteronyssinus and Dermatophagoides farina.

The efficacy of Acarizax has been tested in randomized, double-blinded, placebo-controlled trials as add-on treatment for the best maintenance treatment for AR and AA. The clinical effect of Acarizax has been demonstrated 8-14 weeks after initiation of treatment and data on clinical effect is available for up to 18 months of treatment. Acarizax was found to reduce time to first exacerbation (hazard-ratio 0.7) in patients with AA. Acarizax has been shown to reduce daily mean inhaled corticosteroid (budesonide) by 81 microgram/day (95% CI: 27-136microgram/day). In AR, Acarizax has been shown to reduce Total Combined Rhinitis Score (TCRS). A meta-analysis on the efficacy of AIT on atopic dermatitis shows moderate level of efficacy. Hence, we will be studying the potential change in the immunologic phenotype as an exploratory outcome.

AIT has been known for more than 100 years as a potential curative and specific treatment for allergic diseases. The mechanism by which AIT works is poorly understood but a key target is likely modulation of immunopathology. Dysregulation of the immune system is thought to play an essential role in atopic diseases and is influenced by multiple complex regulatory mechanisms. Well-established immune modulatory effects of AIT are classified into following type of events:

Table 1. Mechanisms of AIT Order of events Events Change Time to initial change

1. Basophil- and Mast cell activity and degranulation of IgE mediated histamine release Decrease Immediately
2. Induction of allergen-specific Treg- and Breg cells and suppression of allergen specific Th1 and Th2 cells Increase Days to weeks
3. Specific IgE Early increase followed by chronic decrease to baseline Weeks to years
4. Specific IgG4 Continuously increase throughout treatment duration Weeks
5. Tissue resident eosinophils, basophils and mast cells and release of their mediators Decrease Months
6. Type 1 skin reactivity decrease Months

1.4 Rationale

Anti-viral immunity Interferons (IFNs) are essential cytokines in the anti-viral defence. IFN's are produced by many cell types in the lungs where human bronchial epithelial cells (HBECs) and plasmacytoid dendritic cells (pDCs) are the main producers. The major effects of IFNs include blocking of viral invasion into neighbour cells by cleaving viral nucleic acid and inhibiting viral replication and inducing apoptosis in affected cells. HBECs are critical for the development of a sufficient innate immune response to viral infection. Increasing evidence suggest that HBECS from patients with asthma and allergic asthma exhibit an impaired ability to secrete type I (IFN-beta), and III (IFN-lambda) interferons at viral infection. In addition, IFN-beta and IFN-lambda may inversely correlate with the level of Type 2 inflammation in the airway epithelium.

pDCs are essential effectors of the primary innate immune defence against viral infections, releasing large amounts of IFN-alpha, and driving Th1 polarisation of CD4 lymphocytes. However, pDCs also play an important role as antigen-presenting cells, by which they may drive a Th2 polarisation, increasing IgE-production in B-cells and potential cross-linking of FcepsilonR1-alpha receptors. Interestingly, it has recently been demonstrated that viral induced IFN-alpha release was diminished by activation of the FcepsilonR1-alpha receptor on the pDC by allergen exposure, suggesting a potential link between allergy and a reduced viral defence. In patients with allergic asthma viral induced IFN-alpha release was impaired in PBMC's indicating a more systemic impact in response to bronchial infection.

AIT: Mechanisms leading to suppression of allergic inflammation In general, it is acknowledged that Th2 / Treg cells tolerance is decisive for the development or suppression of allergic inflammation. Treg cells secrete high amounts of essential suppressor cytokines IL-10 and TGF-beta. These cytokines contribute to the control of Th2 mediated allergic disease in various ways. Treg cells regulates B-cells by inducing a competitive IgG4 and IgA response resulting in suppression of IgE. Furthermore, Treg cells may suppress activation and degranulation of mast cells, basophils and eosinophils. Lastly Treg cells, suppress Th2 cells homing to tissue and epithelial cell activation and production of proinflammatory cytokines. Breg cells control excessive inflammatory responses through secretion of IL-10, supports differentiation of Treg cells and induces synthesis of IgG4. These effects may be involved in response to AIT and correlate with clinical improvement. Thus, AIT may result in a decrease of bronchial, nasal and conjunctival hyperreactivity, which is a reflection of decrease in underlying mucosal inflammation. Anti-IgE treatment ameliorates the seasonal variations in asthma exacerbations associated with virus infections, which may be related to an increase in the initial interferon response to viral infections. We thus speculate, that the potential immunomodulatory effects of AIT resulting in lowered risk of prescription antibiotics is the net result of alteration in allergen-induced mucosal Th-2 inflammation, mediated by an increase in primary IFN defence responses to viral infections.

6.6 Study governance and oversight

6.6.1 Study Site Bispebjerg Hospital, Dep. of Respiratory Medicine Bispebjerg Bakke 23, Entrance 66 DK - 2400 Copenhagen NV Denmark Phone: (+45) 35 31 35 69 Fax: (+45) 35 31 21 79

6.6.12 Additional sites of analyses

* Department of Immunology and Microbiology, University of Copenhagen
* Department of Respiratory Immunopharmacology University of Lund
* ALK-Abelló A/S, Boege Allé 6-8, 2970 Hoersholm

6.6.13 Study registration and authorities Study code: VITAL EudraCT: 2019-003261-18 Ethics Committee journal number: H-19052148 Danish Medicines Agency: 2019-003261-18 ClinicalTrial.gov: NCT04100902

6.6.14 Steering Committee Christian Uggerhoej Woehlk, M.D., Ph.D.-student Asger Sverrild, M.D., Ph.D. Charlotte Menné Bonefeld, Professor Lena Uller Ass. Professor Steen Roenborg, M.D. Ph.D. Celeste Porsbjerg, Professor, M.D.

6.6.15 Participants and collaborators

1. Pharmacy: Region Hovedstadens Apotek, Marielundvej 25, 2730 Herlev, Denmark.
2. Peter Arvidsson, M.D., PhD.: ALK-Abelló Nordic A/S, Kungbacke Sweden
3. Peter Sejer Andersen: ALK-Abelló A/S, Boege Allé 6-8, Bygn. 9, 2970 Hoersholm
4. Peter Adler Würtzen, Senior Specialist, PhD: ALK-Abelló A/S, Boege Allé 6-8, Bygn. 9, 2970 Hoersholm

8. STATISTICAL ANALYSES 8.1 Sample size estimate Sample size calculations have been carried out using G-Power software (Behaviour Research Methods 2007 Faul et al).

8.1.1 Primary outcome:

To our knowledge there is no preceding studies investigation the relationship between AIT treatment and change in IFN-response in HBECS. The investigators have previously shown that treating human airway epithelium in vitro with azithromycin increase the IFN-response to viral infection mimics in a dose-dependent manner. Fold-change in INF-β was 1.55 (SD 0.555) at the given concentration. Given a significant change in IFN-β from week 0 to week 24 is set to be a 1.55-fold change with SD of 0.555, that alpha is set to 0.05, and the power to 0.80, in a two-sided test design, the calculation would look like this:

Mean (fold change in INF-β) group 1 (placebo): 1 Mean (fold change in INF-β) group 2 (Acarizax): 1.55 SD: 0.55 16 subjects will be needed in each study arm. Assuming a drop-out of 20%, a minimum of 40 subjects in total will need to be randomized.

8.2 Definitions of analysis sets 1) Populations for analysis:

1. Intention-to-treat population: All randomized subjects who receive at least one dose of Acarizax or placebo. A comparison of the treatment groups will be performed.

2) Population for analysis based on adherence ≥ 80% to treatment.

1. Intention-to-treat population: All randomized subjects with adherence ≥ 80% to Acarizax therapy or placebo. A comparison of the treatment groups will be performed.

8.2.1 Efficacy analysis set Intention-to-treat population (as defined in 8.2).

8.2.2 Safety analysis set All patients who receive at least one dose of Acarizax/placebo.

8.3 Methods for statistical analyses All data limited to primary and key secondary outcomes will be analysed using SPSS v. 14 or later. all data are reported as median values with interquartile ranges and were analysed using non-parametric tests. Data within each group (Acarizax and placebo) will be analysed using linear mixed model or ANCOVA. Statistical differences between the Acarizax and placebo groups will be determined using the Mann - Whitney U test for unrelated samples. Skewed-data will be log-transformed before analysis and reported using median and 25/75 % percentiles. Parametric data will be analysed using the above-mentioned methods. Categorial data will be analysed using χ²-test. Statistical significance is defined as p<0.05. The data from the subject dropping out will still be used in the analysis using methods for handling of missing data.

8.3.1 Analysis of the primary variable(s) The fold-change in IFN-β and IFN-λ are analysed before and after RV infection and/or poly(I:C) stimulation from V3 to V12 and will be compared between intervention and placebo treatment. The investigators expect parametric distribution of data.

The calculation will be as follows:

1. deltaIFN-β: IFN-β V12 - IFN-βV3
2. Mean fold-change IFN-β: Sum of individual changes / N

Supportive primary objectives are calculated between intervention and placebo treatment groups:

1. Change in expression of IFN-λ measured in ρg/ml (ELISA) and reported as fold change mean ± SD
2. Change in viral load/TCID50 assay measure reported as fold change mean ± SD

8.3.2 Analysis of the secondary variable(s)

* Changes in IFN-responses will be analysed using same procedure as analysis of the primary outcome.
* Cytokines will be analysed accordingly to the method described in 8.3.1 and reported as ρm/ml (or similar quantitative method) and reported as fold change mean ± SEM
* Change in IFN-β/TSLP ratio and reported in %.
* The change, expressed as a ratio, in number of airway submucosal, muscle and epithelium mast cells, eosinophils, neutrophils, NK-cells, (MCT, MCTC and MCCPA3) per mm2 determined by microscopic evaluation of mucosa biopsies and epithelial brushings from V2 to V7.

8.3.3 Interim analysis No interim analysis is planned.

8.3.4 Use of database REDCap will be used for online CRF data management.

9. STUDY AND DATAMANGEMENT 9.1 Economy

The scientific ideas of protocol are based solely on the work of members of the steering committee. None of the members of the steering committee have any commercial interest in the results of this study. As per 01.08.19, the project has received:

1. Unrestricted grant from ALK-Abelló Nordic of (900.000dkk)
2. Unrestricted grant from Sawmill owner Jeppe Juhl and wife Ovita Juhls memorial fund (250.000 dkk).
3. HARBOEFONDEN: DKK 200.000
4. Pharmaxis: Osmohale Mannitol Challenge tests

9.2. Subject reimbursement Each subject completing the study will receive a total of 6 months of Acarizax treatment equivalent to approximate 5.500 dkk. Subject randomized to Acarizax arm will not be furtherly compensated.

9.2.1 Source data Will be filed at Bispebjerg Hospital, Denmark (study site) in accordance with The Danish Data Protection Agency laws. Source data will be kept for a maximum of 20 years from (01.09.2019). At this point all source data will be destroyed.

9.2.2 Study agreements All agreements relating to the study will be available in the trial master file (TMF).

9.2.3 Archiving of study documents Documents will be archived at Bispebjerg Hospital, Denmark (study site) in accordance with GCP and The Danish Data Protection Agency laws.

9.3 Monitoring of the study

The study will be monitored by the GCP Unit in Copenhagen:

Copenhagen University Hospital GCP-unit Bispebjerg Hospital, Building 51, 3.fl Bispebjerg Bakke 23 DK - 2400 København NV Denmark Phone: (+45) 3531 3887 E-mail: gcp-enheden.bispebjerg-frederiksberg-hospitaler@regionh.dk www.gcp-enhed.dk.

ELIGIBILITY:
Subjects must meet all the following criteria:

INCLUSION CRITERIA

1. Written informed consent
2. Age ≥18 through ≤ 65, inclusive at the time of V1
3. A historic verified diagnosis of asthma as defined by 1 positive of following tests:

   1. Reversibility to Beta-2-agonist
   2. Positive mannitol challenge test
   3. Positive methacholine test
   4. Positive peak-flow variation test
   5. Positive eucapnic voluntary hyperventilation test
   6. Exercise test
4. Mild to severe symptoms of of HDM induced rhinitis for at least one year (acc. ARIA 2008 Bousqet et al. 2008).
5. ≥1 self-reported worsening of asthma symptoms in relations to viral infection within last 12 months

7. A postbronchodilator FEV1 value of ≥ 70% at V1

8. ACQ-6 ≥ 1 at V1

9. A stable asthma controller regimen with ICS for at least 4 weeks prior to V1 (GINA 2-4)

10. Daily dose of ICS at V1 (budesonide equivalent) ≥400µg 11. Sensitisation to HDM defined by one of the following:

1. Positive skin prick test defined as a wheel diameter ≥ 3 mm for either: Dermatophagoides pteronyssinus or Dermatophagoides farina

   OR
2. IgEHDM > 0.7 x103 IU/L

   12. Subjects must demonstrate acceptable inhaler and spirometry techniques during screening (as evaluated and in the opinion of study site staff)

EXCLUSION CRITERIA

Any of the following would exclude the subject from participation in the study:

1. Oral corticosteroids (any dose for more than 3 days) 8 weeks prior to V1 and during run-in.
2. Acute upper or lower respiratory infections requiring antibiotics or antiviral medications 6 weeks prior to V1 and during run-in.
3. Severe oral conditions such as but not limited to:

   1. Oral ulcers
   2. Oral lichen planus
   3. Oral mycosis
4. Smoking any kind

   1. Quit > 6 months prior to V1.
   2. ≥ 10 pack years
5. Positive skin prick test defined as a wheel diameter ≥ 3 mm:

   a. Alternaria, Cladosporium, Aspergillus
6. Positive skin prick test defined as a wheel diameter ≥ 3 mm for- and with anamnestic relevant exposure to:

   a. Cat, Dog, Horse
7. Ever in treatment with any AIT
8. Previous medical history or evidence of an uncontrolled intercurrent illness such as but not limited to (e.g. Autoimmune disease, immunodeficiency, immunosuppression, malignant neoplastic conditions with current relevance) that in the opinion of the investigator may compromise the safety of the subject in the study or interfere with evaluation of the investigational product or reduce the subject's ability to participate in the study. Subjects with well-controlled comorbid disease (eg, hypertension, hyperlipidaemia, gastroesophageal reflux disease) on a stable treatment regimen for 15 days prior to V1 are eligible.
9. Any concomitant respiratory disease that in the opinion of the investigator and/or medical monitor will interfere with the evaluation of the investigational product or interpretation of subject safety or study results (eg, chronic obstructive pulmonary disease, cystic fibrosis, pulmonary fibrosis, bronchiectasis, allergic bronchopulmonary aspergillosis, Churg-Strauss syndrome, alpha-1-antitrypsin deficiency, Wegeners granulomatosis, Sarcoidosis).
10. Any clinically relevant abnormal findings in haematology or clinical chemistry (laboratory results from Visit 1), physical examination, vital signs during the screening, which in the opinion of the investigator, may put the subject at risk because of his/her participation in the study, or may influence the results of the study, or the subject's ability to participate in the study.
11. Evidence of active liver disease, including jaundice, alanine transaminase, bilirubin, greater than twice the upper limit of normal (laboratory results from V1).
12. History of cancer:

    1. Subjects who have had basal cell carcinoma or in situ carcinoma of the cervix are eligible to participate in the study provided that curative therapy was completed at least 12 months prior to V1.
    2. Subjects who have had other malignancies are eligible provided that curative therapy was completed at least 5 years prior to V1.
13. A helminth parasitic infection diagnosed within 24 weeks of V1 that has not been treated or has not responded to standard of care therapy.
14. Known history of active tuberculosis (TB). Subjects may be enrolled if they have ALL of the following:

    1. No symptoms of TB: productive, prolonged cough (> 3 weeks); coughing up blood; fever; night sweats; unexplained appetite loss; unintentional weight loss.
    2. No known exposure to a case of active TB after most recent prophylaxis (prophylaxis required only if positive).
    3. No evidence of active TB on chest radiograph within 3 months prior to the first dose of investigational product.
15. Positive hepatitis B surface antigen, or hepatitis C virus antibody serology at screening, or a positive medical history for hepatitis B or C. Subjects with a history of hepatitis B vaccination without history of hepatitis B are allowed to enrol.
16. A positive human immunodeficiency virus (HIV) test at screening or subject taking antiretroviral medications, as determined by medical history and/or subject's verbal report.
17. History of any known primary immunodeficiency disorder excluding asymptomatic selective immunoglobulin A or IgG subclass deficiency.
18. Use of 5-lipoxygenase inhibitors (eg, zileuton) within 15 days prior to V1.
19. Use of immunosuppressive medication (eg, methotrexate, troleandomycin, oral gold, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroid, or any experimental anti-inflammatory therapy) within 3 months prior to V1.
20. Receipt of any of the following within 30 days prior to V1:

    1. Immunoglobulin or blood products, or
    2. Receipt of any investigational nonbiologic agent within 30 days or 5 half-lives prior Visit 1, whichever is longer.
21. Receipt or treatment with of any marketed or investigational biologic agent within 6 months or 5 half-lives prior to V1, whichever is longer, specifically:

    1. Anti-IgE
    2. Anti-IL4
    3. Anti-IL-5
    4. Anti-IL5 receptor antagonist
    5. Anti-IL-13
22. Pregnant, breastfeeding or lactating females
23. History of chronic alcohol or drug abuse within 12 months prior to V1.
24. Planned surgical procedures requiring general anaesthesia or in-patient status for > 1 day during the conduct of the study.
25. Unwillingness or inability to follow the procedures outlined in the protocol.
26. Concurrent enrolment in another clinical study involving an investigational treatment.
27. Receipt of the Th2 cytokine inhibitor Suplatast Tosilate within 15 days prior to V1.
28. Receipt of any live or attenuated vaccines within 15 days prior to V1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
ΔIFN-ß gene and/or protein expression | Baseline and 24 weeks
  To investigate the potential change in viral induced interferon response in HBECs from V3, V12, after 24 weeks of HDM-SLIT therapy or placebo, after stimulation with a combination of: HDM-allergen +/- viral infection mimics (RV16 or Poly(I:C))
ΔIFN-λ gene and/or protein expression | Baseline and 24 weeks
  To investigate the potential change in viral induced interferon response in HBECs from V3, V12, after 24 weeks of HDM-SLIT therapy or placebo, after stimulation with a combination of: HDM-allergen +/- viral infection mimics (RV16 or Poly(I:C))
ΔViral load | Baseline and 24 weeks
  To investigate the potential change in viral load in HBECS from from V3, V12, after 24 weeks of HDM-SLIT therapy or placebo, after stimulation with a combination of HDM-allergen +/- viral infection mimics (RV16 or Poly(I:C))

SECONDARY OUTCOMES:
ΔIFN-ß gene and/or protein expression in viral/bacterial co-stimulation assay | Baseline and 24 weeks
  To investigate the potential change in viral induced interferon response in HBECs from V3 to V12, after 24 weeks of HDM-SLIT therapy, after stimulation with a combination of: HDM-allergen +/- viral infection mimics (RV16 or Poly(I:C) +/- bacterial infection mimics
ΔIFN-λ gene and/or protein expression in viral/bacterial co-stimulation assay | Baseline and 24 weeks
  To investigate the potential change in viral induced interferon response in HBECs from V3 to V12, after 24 weeks of HDM-SLIT therapy, after stimulation with a combination of: HDM-allergen +/- viral infection mimics (RV16 or Poly(I:C) +/- bacterial infection mimics
ΔIL-12 | Baseline and 24 weeks
  To investigate the potential change in IL-12 response in HBECs from V3 to V12, after 24 weeks of HDM-SLIT therapy, after stimulation with a combination of: HDM-allergen +/- viral infection mimics (RV16 or Poly(I:C) +/- bacterial infection mimics
Δß-defensin | Baseline and 24 weeks
  To investigate the potential change in ß-defensin response in HBECs from V3 to V12, after 24 weeks of HDM-SLIT therapy, after stimulation with a combination of: HDM-allergen +/- viral infection mimics (RV16 or Poly(I:C) +/- bacterial infection mimics
ΔIFN-γ | Baseline and 24 weeks
  To investigate the potential change in IFN- γ response in HBECs from V3 to V12, after 24 weeks of HDM-SLIT therapy, after stimulation with a combination of: HDM-allergen +/- viral infection mimics (RV16 or Poly(I:C) +/- bacterial infection mimics
Th1/Th2 balance | Baseline and 24 weeks
  To investigate the potential change in immunologic phenotype in BAL-fluid from V3 to V12, after 24 weeks of HDM-SLIT therapy. Analyses will be performed using flowcytometri and/or ELISA/Luminex/MSD
ΔNK-cells | Baseline and 24 weeks
  To investigate the potential change in immunologic phenotype in BAL-fluid from V3 to V12, after 24 weeks of HDM-SLIT therapy. Analyses will be performed using flowcytometri and/or ELISA/Luminex/MSD
ΔCD8+ T-cells. | Baseline and 24 weeks
  To investigate the potential change in immunologic phenotype in BAL-fluid from V3 to V12, after 24 weeks of HDM-SLIT therapy. Analyses will be performed using flowcytometri and/or ELISA/Luminex/MSD
Inflammatory cytokines such as but not restricted to: IL-4, IL-5, IL-13, IL-33, IL-25, IL-ß and TSLP | Baseline and 24 weeks
  To investigate the potential change in immunologic phenotype in BAL-fluid from V3 to V12, after 24 weeks of HDM-SLIT therapy. Analyses will be performed using flowcytometri and/or ELISA/Luminex/MSD
IFN-ß/TSLP ratio | Baseline and 24 weeks
  To investigate the potential change in the cell supernatants for epithelial derived Th1/Th2-cytokines as well as Th1/Th2 (anti)-inflammatory cytokines.
Mast cells, eosinophils, Neutrophils, pDC's | Baseline and 24 weeks
  To evaluate the potential change in histologic phenotype in bronchial biopsies from V3 to V12, after 24 weeks of HDM-SLIT therapy
Number / percentage of eosinophils and neutrophils in sputum. | Baseline and 24 weeks
  To investigate potential change in airway inflammation markers in sputum
IFN-ß(λ)/SOCS1/(3)-ratio | Baseline and 24 weeks
  To investigate potential invers relation between IFN production and SOCS1 expression
IFN-ß(λ)/TLR3(7)-ratio | Baseline and 24 weeks
  To investigate potential invers relation between IFN production and SOCS1
SOCS 1 immunohistochemistry. | Baseline and 24 weeks
  Expression of SOCS 1 in nucleus in bronchial biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Porsbjerg, Professor, Principal Investigator — Respiratory Research Unit, department of Respiratory Medicine, Bispebjerg University Hospital
Locations (1):
- Respiratory Research Unit, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woehlk C, Ramu S, Sverrild A, Nieto-Fontarigo JJ, Vazquez-Mera S, Cerps S, Pulga A, Andreasson LM, Eriksen LL, Dyhre-Petersen N, Menzel M, Klein DK, Hansen S, Uller L, Porsbjerg C. Allergen Immunotherapy Enhances Airway Epithelial Antiviral Immunity in Patients with Allergic Asthma (VITAL Study): A Double-Blind Randomized Controlled Trial. Am J Respir Crit Care Med. 2023 May 1;207(9):1161-1170. doi: 10.1164/rccm.202209-1708OC. PMID 36701676